CLINICAL TRIAL: NCT01165242
Title: Immunogenicity and Safety Study of One Dose of GSK Biologicals' Meningococcal Vaccine GSK 134612 (Blinded Lots) Versus One Dose of Menactra® in Healthy Subjects Aged 10-25 Years
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' Meningococcal Vaccine GSK 134612 Versus Menactra® in Healthy Adolescents/Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 114249
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Infections, Meningococcal
Keywords: Neisseria meningitidis; Adult; Adolescent; Safety; Vaccines, conjugate; Meningococcal vaccines; Immunogenicity
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Group A (Experimental): Subjects were vaccinated with vaccine GSK134612 Lot A
  Interventions: Biological: Meningococcal vaccine GSK 134612
- Group B (Experimental): Subjects were vaccinated with vaccine GSK134612 Lot B
  Interventions: Biological: Meningococcal vaccine GSK 134612
- Group C (Active Comparator): Subjects were vaccinated with Menactra®
  Interventions: Biological: Menactra®

INTERVENTIONS:
Biological: Meningococcal vaccine GSK 134612 — One intramuscular injection
  Arms: Group A; Group B
Biological: Menactra® — One intramuscular injection
  Arms: Group C

SUMMARY:
The purpose of this observer-blind study is to evaluate the safety and immunogenicity of GSK Biologicals' meningococcal vaccine GSK134612 as compared to Menactra® in subjects 10 through 25 years of age. In addition, this study will compare the immunogenicity of two lots of GSK 134612 vaccine.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL of the following criteria at study entry:

* Subjects whom the investigator believes that they and/or their parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* A male or female between, and including, 10 and 25 years of age at the time of the vaccination.
* Written informed consent obtained from the subject/from the parent or Legally Acceptable Representative(s) of the subject. Assent will be obtained from subjects who are still legally minors in line with local rules and regulations.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of subject's/Legally Acceptable Representative(s)'s knowledge.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception for 2 months after vaccination.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to vaccination. (For corticosteroids, this will mean prednisone <10 mg/day, or equivalent, is allowed. Inhaled and topical steroids are allowed.)
* Planned administration/administration of a vaccine not foreseen by the study protocol within one month of the dose of vaccine, with the exception of any licensed inactivated influenza vaccine.
* Previous vaccination with meningococcal polysaccharide or conjugate vaccine.
* Previous vaccination with vaccine components within the last month.
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of allergic reactions or disease likely to be exacerbated by any component of either vaccine, or by dry natural rubber latex.
* History of any neurologic disorders, including Guillain-Barré Syndrome.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrollment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy.
* Child in care.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1013 (Actual)
Dates: Start 2010-08-19; Primary Completion 2011-02-25 (Actual); Study Completion 2011-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (22):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Nicholasville, Kentucky
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Albany, Oregon
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Austin, Texas
- Canada (8):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Halperin SA, Baine Y, Domachowske JB, Aggarwal N, Simon M, Langley JM, McNeil SA, Friedland LR, Bianco V, Baccarini CI, Miller JM. Comparison of the Safety and Immunogenicity of a Novel Quadrivalent Meningococcal ACWY-Tetanus Toxoid Conjugate Vaccine and a Marketed Quadrivalent Meningococcal ACWY-Diphtheria Toxoid Conjugate Vaccine in Healthy Individuals 10-25 Years of Age. J Pediatric Infect Dis Soc. 2014 Mar;3(1):33-42. doi: 10.1093/jpids/pit058. Epub 2013 Oct 17. PMID 24567843
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114249 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 1013 subjects enrolled in this study, 2 were assigned subject numbers but received no vaccination and were hence excluded from the study start.
Groups:
- Nimenrix Lot A Group: Healthy male and female subjects between, and including, 10 and 25 years of age, who received 1 dose of Nimenrix Lot A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
- Nimenrix Lot B Group: Healthy male and female subjects between, and including, 10 and 25 years of age, who received 1 dose of Nimenrix Lot B vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
- Menactra Group: Healthy male and female subjects between, and including, 10 and 25 years of age, who received 1 dose of Menactra vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
Started | 337 | 336 | 338
Completed | 327 | 326 | 324
Not Completed | 10 | 10 | 14
Not completed — Unreachable Subjects | 1 | 0 | 0
Not completed — Incarcerated Subjects | 0 | 1 | 0
Not completed — Visit 2 Declined by Subject | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Extended Holiday | 0 | 0 | 1
Not completed — Lost to Follow-up | 9 | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group | Total
Number analyzed (Participants) | 337 | 336 | 338 | 1011
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.4 (5.16) | 16.3 (5.16) | 16.2 (4.97) | 16.30 (5.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 169 | 176 | 520
  Male | 162 | 167 | 162 | 491
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage/ African American | 38 | 29 | 40 | 107
  Geographic ancestry: American Indian or Alaskan Native | 4 | 2 | 1 | 7
  Geographic ancestry: Asian-Central/ South Asian Heritage | 17 | 17 | 17 | 51
  Geographic ancestry: Asian - East Asian Heritage | 4 | 3 | 5 | 12
  Geographic ancestry: Asian - Japanese Heritage | 0 | 2 | 0 | 2
  Geographic ancestry: Asian - South East Asian Heritage | 4 | 3 | 2 | 9
  Geographic ancestry: White - Arabic/ North African Heritage | 2 | 3 | 2 | 7
  Geographic ancestry: White - Caucasian/ European Heritage | 248 | 249 | 257 | 754
  Geographic ancestry: Other (Mix of races, e.g. African/White) | 20 | 28 | 14 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Response to Serum Bactericidal Assay Using Human Complement Against Neisseria Meningitidis Serogroup A, C, W-135 and Y (hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY) Antibodies
Description: Vaccine response was defined as:
  * for initially seronegative subjects [with hSBA titer below (<) 1:4]: post-vaccination antibody titer greater than or equal to (≥) 1:8 one month after vaccination;
  * for initially seropositive subjects (with hSBA titer ≥ 1:4): post-vaccination antibody titer ≥ 4-fold the pre-vaccination antibody titer one month after vaccination.
Time Frame: One month after vaccination (Month 1)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who had received the study vaccine dose and for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Lot A Group | Menactra Group
Number analyzed (Participants) | 310 | 297
Participants
  hSBA-MenA | 218 | 191
  hSBA-MenC: number analyzed (Participants) | 281 | 274
  hSBA-MenC | 217 | 209
  hSBA-MenW-135: number analyzed (Participants) | 279 | 289
  hSBA-MenW-135 | 198 | 185
  hSBA-MenY: number analyzed (Participants) | 293 | 295
  hSBA-MenY | 150 | 115

2. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the hSBA-Men titers was greater than or equal to (≥) 1:4.
Time Frame: Prior to (PRE) and one month after vaccination (Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who had received the study vaccine dose and for whom assay results were available for antibodies against at least one study vaccine antigen component.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
Number analyzed (Participants) | 315 | 309 | 306
Participants
  hSBA-MenA, PRE: number analyzed (Participants) | 310 | 309 | 306
  hSBA-MenA, PRE | 79 | 84 | 89
  hSBA-MenA, Month 1: number analyzed (Participants) | 315 | 309 | 305
  hSBA-MenA, Month 1 | 253 | 243 | 223
  hSBA-MenC, PRE: number analyzed (Participants) | 288 | 286 | 289
  hSBA-MenC, PRE | 175 | 188 | 197
  hSBA-MenC, Month 1: number analyzed (Participants) | 307 | 304 | 296
  hSBA-MenC, Month 1 | 295 | 293 | 291
  hSBA-MenW-135, PRE: number analyzed (Participants) | 293 | 290 | 299
  hSBA-MenW-135, PRE | 99 | 98 | 102
  hSBA-MenW-135, Month 1: number analyzed (Participants) | 298 | 292 | 297
  hSBA-MenW-135, Month 1 | 272 | 262 | 247
  hSBA-MenY, PRE: number analyzed (Participants) | 296 | 306 | 304
  hSBA-MenY, PRE | 215 | 224 | 234
  hSBA-MenY, Month 1: number analyzed (Participants) | 313 | 307 | 305
  hSBA-MenY, Month 1 | 307 | 302 | 287

3. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for the hSBA-Men titers was greater than or equal to (≥) 1:8.
Time Frame: Prior to (PRE) and one month after vaccination (Month 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
Number analyzed (Participants) | 315 | 309 | 306
Participants
  hSBA-MenA, PRE: number analyzed (Participants) | 310 | 309 | 306
  hSBA-MenA, PRE | 61 | 65 | 67
  hSBA-MenA, Month 1: number analyzed (Participants) | 315 | 309 | 305
  hSBA-MenA, Month 1 | 251 | 242 | 221
  hSBA-MenC, PRE: number analyzed (Participants) | 288 | 286 | 289
  hSBA-MenC, PRE | 174 | 185 | 193
  hSBA-MenC, Month 1: number analyzed (Participants) | 307 | 304 | 296
  hSBA-MenC, Month 1 | 295 | 292 | 291
  hSBA-MenW-135, PRE: number analyzed (Participants) | 293 | 290 | 299
  hSBA-MenW-135, PRE | 99 | 97 | 101
  hSBA-MenW-135, Month 1: number analyzed (Participants) | 298 | 292 | 297
  hSBA-MenW-135, Month 1 | 272 | 262 | 247
  hSBA-MenY, PRE: number analyzed (Participants) | 296 | 306 | 304
  hSBA-MenY, PRE | 215 | 223 | 234
  hSBA-MenY, Month 1: number analyzed (Participants) | 313 | 307 | 305
  hSBA-MenY, Month 1 | 307 | 302 | 287

4. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to (PRE) and one month after vaccination (Month 1)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
Number analyzed (Participants) | 315 | 309 | 306
Titers
  hSBA-MenA, PRE: number analyzed (Participants) | 310 | 309 | 306
  hSBA-MenA, PRE | 3.6 [3.1 to 4.0] | 3.6 [3.2 to 4.1] | 3.6 [3.2 to 4.1]
  hSBA-MenA, Month 1: number analyzed (Participants) | 315 | 309 | 305
  hSBA-MenA, Month 1 | 54.2 [43.5 to 67.4] | 49.6 [39.6 to 62.1] | 41.3 [32.3 to 52.9]
  hSBA-MenC, PRE: number analyzed (Participants) | 288 | 286 | 289
  hSBA-MenC, PRE | 15.6 [12.3 to 19.9] | 16.0 [12.8 to 20.0] | 18.0 [14.4 to 22.6]
  hSBA-MenC, Month 1: number analyzed (Participants) | 307 | 304 | 296
  hSBA-MenC, Month 1 | 687.1 [510.5 to 924.9] | 755.8 [557.3 to 1025.0] | 543.3 [411.2 to 718.0]
  hSBA-MenW-135, PRE: number analyzed (Participants) | 293 | 290 | 299
  hSBA-MenW-135, PRE | 7.7 [6.1 to 9.7] | 7.6 [6.0 to 9.6] | 7.4 [5.9 to 9.2]
  hSBA-MenW-135, Month 1: number analyzed (Participants) | 298 | 292 | 297
  hSBA-MenW-135, Month 1 | 174.5 [138.6 to 219.6] | 161.6 [128.3 to 203.5] | 101.7 [77.9 to 132.7]
  hSBA-MenY, PRE: number analyzed (Participants) | 296 | 306 | 304
  hSBA-MenY, PRE | 45.7 [35.9 to 58.2] | 49.8 [39.1 to 63.4] | 55.3 [43.7 to 69.9]
  hSBA-MenY, Month 1: number analyzed (Participants) | 313 | 307 | 305
  hSBA-MenY, Month 1 | 349.1 [298.1 to 408.8] | 387.4 [329.7 to 455.1] | 253.8 [204.9 to 314.5]

5. Secondary Outcome: Number of Subjects With Vaccine Response for hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibodies
Description: Vaccine response was defined as: -for initially seronegative subjects [with hSBA titer below (<) 1:4]: post-vaccination antibody titer greater than or equal to (≥) 1:8 one month after vaccination; -for initially seropositive subjects (with hSBA titer ≥ 1:4): post-vaccination antibody titer ≥ 4-fold the pre-vaccination antibody titer one month after vaccination.
Time Frame: One month after vaccination (Month 1)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who had received the study vaccine dose and for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Lot B Group
Number analyzed (Participants) | 300
Participants
  hSBA-MenA | 214
  hSBA-MenC: number analyzed (Participants) | 274
  hSBA-MenC | 226
  hSBA-MenW-135: number analyzed (Participants) | 270
  hSBA-MenW-135 | 196
  hSBA-MenY: number analyzed (Participants) | 294
  hSBA-MenY | 150

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
Number analyzed (Participants) | 329 | 329 | 325
Participants
  Any Pain | 169 | 167 | 180
  Grade 3 Pain | 8 | 5 | 2
  Any Redness | 85 | 60 | 66
  Grade 3 Redness | 3 | 2 | 6
  Any Swelling | 63 | 40 | 44
  Grade 3 Swelling | 3 | 3 | 3

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal, headache and temperature [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
Number analyzed (Participants) | 329 | 329 | 326
Participants
  Any Fatigue | 96 | 94 | 89
  Grade 3 Fatigue | 9 | 7 | 5
  Related Fatigue | 75 | 80 | 77
  Any Gastrointestinal | 43 | 43 | 44
  Grade 3 Gastrointestinal | 4 | 3 | 4
  Related Gastrointestinal | 31 | 33 | 32
  Any Headache | 86 | 87 | 83
  Grade 3 Headache | 5 | 2 | 6
  Related Headache | 72 | 70 | 68
  Any Temperature (Orally) | 17 | 14 | 16
  Grade 3 Temperature (Orally) | 1 | 0 | 0
  Related Temperature (Orally) | 15 | 10 | 12

8. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (Day 0-30) post-vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
Number analyzed (Participants) | 337 | 336 | 338
Participants | 105 | 76 | 85

9. Secondary Outcome: Number of Subjects With New Onset of Chronic Illness(es) (NOCI)
Description: NOCI included hypersensitivity, insulin resistance, asthma and bronchial hyperreactivity.
Time Frame: From Month 0 through Month 6
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
Number analyzed (Participants) | 337 | 336 | 338
Participants | 3 | 0 | 0

10. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 through Month 6
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
Number analyzed (Participants) | 337 | 336 | 338
Participants | 1 | 5 | 2

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period. Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period. SAEs: during the entire study period (from Month 0 up to Month 6).
Description: The solicited local and general symptoms were only collected from those subjects who filled in their symptom sheets.
Arm/Group | Nimenrix Lot A Group | Nimenrix Lot B Group | Menactra Group
All-Cause Mortality (participants affected / at risk) | 0/337 | 0/336 | 0/338
Serious Adverse Events (participants affected / at risk) | 1/337 | 5/336 | 2/338
Other Adverse Events (participants affected / at risk) | 232/337 | 219/336 | 234/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix Lot A Group (N=337) | Nimenrix Lot B Group (N=336) | Menactra Group (N=338)
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix Lot A Group (N=337) | Nimenrix Lot B Group (N=336) | Menactra Group (N=338)
Pain (General disorders) | 169/329 | 167/329 | 180/325 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Redness (General disorders) | 85/329 | 60/329 | 66/325 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Swelling (General disorders) | 63/329 | 40/329 | 44/325 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Fatigue (General disorders) | 96/329 | 94/329 | 89/326 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Gastrointestinal (General disorders) | 43/329 | 43/329 | 44/326 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Headache (General disorders) | 86/329 | 87/329 | 83/326 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Temperature (Orally) (General disorders) | 17/329 | 14/329 | 16/326 — This solicited general symptom was only collected from subjects with their symptom sheets completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.